CLINICAL TRIAL: NCT05441514
Title: Phase 1b Study of IDH Inhibition With Enasidenib and MEK Inhibition With Cobimetinib in Patients With Relapsed or Refractory Acute Myeloid Leukemia Who Have Co-Occurring IDH2 and RAS Signaling Gene Mutations
Brief Title: Enasidenib in Combination With Cobimetinib for the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21751; NCI-2022-04926 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21751 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cobimetinib; 2-Propanol; methanesulfonic acid; enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cobimetinib, enasidenib mesylate) (Experimental): Patients receive cobimetinib PO QD on days 1-21 and enasidenib mesylate PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cobimetinib; Drug: Enasidenib Mesylate

INTERVENTIONS:
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
Drug: Enasidenib Mesylate — Given PO
  Other Names: 2-Methyl-1-[(4-[6-(trifluoromethyl)pyridin-2-yl]-6-{[2-(trifluoromethyl)pyridin-4-yl]amino}-1,3,5-triazin-2-yl)amino]propan-2-ol Methanesulfonate; 2-Propanol, 2-Methyl-1-((4-(6-(trifluoromethyl)-2-pyridinyl)-6-((2-(trifluoromethyl)-4-pyridinyl)amino)-1,3,5-triazin-2-yl)amino)-, Methanesulfonate (1:1); AG-221 Mesylate; CC-90007; Enasidenib Methanesulfonate; Idhifa

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of a enasidenib in combination with cobimetinib in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). Enasidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Cobimetinib is used in patients whose cancer has a mutated (changed) form of a gene called BRAF. It is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Giving enasidenib and cobimetinib may kill more cancer cells in patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of cobimetinib in combination with enasidenib.

II. Determine the maximum tolerated dose(s) (MTD) and recommended phase 2 dose (RP2D).

SECONDARY OBJECTIVES:

I. Obtain preliminary estimates of clinical activity as measured by the complete remission (complete response [CR], complete response with incomplete hematologic recovery [CRi], or complete response with partial hematologic recovery [CRh]) rate and minimal residual disease (MRD) rate.

II. Obtain preliminary estimates of clinical activity as measured by overall response rate (CR, CRi, CRh, morphologic leukemia free state [MLFS], and partial response [PR]).

III. Obtain preliminary estimates of median time to complete remission. IV. Obtain preliminary estimates of median time to first response. V. Obtain preliminary estimates of response duration in all participants and in those attaining CR/CRi/CRh.

VI. Obtain preliminary estimates of median and 1-year event-free survival (EFS).

VII. Obtain preliminary estimates of median and 1-year overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Characterize the effects of the combination on cellular differentiation of leukemic cells as measured by flow cytometry performed at study entry and at serial timepoints throughout the study.

II. Evaluate changes in promotor methylation patterns after treatment with combination therapy.

III. Evaluate changes in gene expression of RAS pathway regulators as a result of the combination therapy.

OUTLINE: This is dose-escalation study of cobimetinib followed by a dose-expansion study.

Patients receive cobimetinib orally (PO) once daily (QD) on days 1-21 and enasidenib mesylate PO QD on days 1-28 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and every 3 months for 1 year at last treatment dose.

ELIGIBILITY:
Main Inclusion Criteria

* Patients with histologically confirmed AML, according to WHO criteria, with refractory/relapsed (R/R) disease who are ineligible for therapies known to be effective for treatment of their AML.

  * Patients with non-central nervous system (CNS) extramedullary disease may be included if they also have marrow involvement
  * Patients with acute promyelocytic leukemia (APL) will not be eligible
  * Patients with IDH2 mutations, who were previously treated with enasidenib are allowed
* Have a documented IDH2 gene mutation (≥ 2% allele frequency) and a concomitant detectable RAS-pathway mutation (as determined by local testing), involving NRAS, KRAS, HRAS, BRAF, KIT, RIT1, PTPN11, CBL or NF1 genes.
* Adults aged ≥ 18 years
* ECOG ≤ 2
* WBC ≤25 x 10^9/L prior to initiation of enasidenib.

Main Exclusion Criteria

* Current or planned use of other investigational agents, antineoplastic, chemotherapy, radiation therapy, biological therapy, immunotherapy or major surgery within 2 weeks or 5 half-lives, whichever is shorter, prior to Day 1 of protocol therapy (exception: hydroxyurea is allowed in cycles 1 and 2 for control of rapidly progressing leukemia or for treatment of enasidenib-related leukocytosis)
* Systemic steroid therapy > 10 mg/day (≤ 10mg/day prednisone equivalent ok) or any other form of immunosuppressive medication within 28 days, except as required for treatment of differentiation syndrome
* Strong and moderate CYP3A4 inducers/inhibitors (moderate CYP3A4 inhibitors only allowed on Principal Investigator approval) within 14 days or 5 half-lives, whichever is shorter, prior to Day 1 of protocol therapy
* Foods/supplements that are strong or moderate inhibitors or inducers of CYP3A (such as grapefruit, Seville oranges, starfruit and St. John's wort) within 7 days prior to initiation of and during study treatment
* Gastrointestinal disorder such as maladsorption syndrome or any other disorder that may interfere with oral drug absorption
* Clinically significant cardiac morbidities (Class III/IV cardiovascular disability according to the New York Heart Association Classification, arrhythmia not stable on medical management, acute cardiovascular ischemic event within 6 months of enrollment, etc)
* Active CNS disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Cycle 1 (28 days)
  Toxicity will be graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Incidence of adverse events | Up to 30 days after last dose of study drug
  Toxicity will be graded according to the NCI- CTCAE version 5.0. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Response | Up to 1 year
  Response will be determined using European LeukemiaNet (ELN) criteria.
Minimal residual disease (MRD) status | Up to 1 year
  MRD status will be determined by standard of care (SOC) flow cytometry assay.
Complete remission | Up to 1 year
  Time to complete remission is defined as time from first study dose to attainment of complete response(CR), complete response with incomplete hematologic recovery CRi, or complete response with partial hematologic recovery CRh). Will calculate rates and 95% Clopper-Pearson binomial confidence interval (CI).
Time to first response | From first study does to first documented complete response, assessed up to 3 years
  Time to first response is defined as time from first study dose to attainment of first documented CR, CRi, CRh, morphologic leukemia free state (MLFS), or partial response (PR). Will calculate rates and 95% Clopper-Pearson binomial CI.
Response duration | From first study does to first documented complete response, assessed up to 1 year
  Response Duration is defined as the time from the date of first documented response (CR, CRi, CRh, MLFS or PR) to documented disease relapse/progression or death, whichever occurs first. Will be estimated using the product-limit method of Kaplan and Meier.
Event-free survival (EFS) | From first study dose to first documented complete response to relapse/progression (> 5% blasts, reappearance of blasts in blood, or development of extramedullary disease) or death, whichever occurs first, assessed up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.
Overall survival (OS) | From first study dose to death from any cause, assessed up to 1 year
  Will be estimated using the product-limit method of Kaplan and Meier.

OTHER OUTCOMES:
Level of myeloid differentiation | Up to 1 year
  Level of myeloid differentiation on pre and post-treatment peripheral blood (PB) and bone marrow (BM) samples by flow cytometry.
Promotor methylation status of RAS pathway regulator | Up to 1 year
  Promotor methylation status of RAS pathway regulators by enhanced reduced representation bisulfite sequencing.
Changes in RAS pathway regulatory gene expression levels | Pre and post- treatment, assessed up to 1 year
  Changes in RAS pathway regulatory gene expression levels by ribonucleic acid (RNA) sequencing pre- and post-treatment. Will use Next generation sequencing (HopeSeq) and/or rapid sequencing assays (Rapid AML Panel).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ball, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States